CLINICAL TRIAL: NCT05413824
Title: Neutrophil Side Fluorescent Light (NEU-SFL) in COVID-19 Patients Hospitalized in 2021
Brief Title: Neutrophil Side Fluorescent Light (NEU-SFL) in COVID-19 Patients
Acronym: NEU-COVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2022/SB-01
Record Dates: First submitted 2022-06-09; First posted 2022-06-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: COVID-19; neutrophil extracellular traps (NETs)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 survivors: Patients hospitalized at Nimes university hospital in 2021 for COVID-19 who survived.
- COVID-19 Deceased: Patients hospitalized at Nimes university hospital in 2021 for COVID-19 who died.

SUMMARY:
Recently, a study showed that markers of neutrophil extracellular traps formation, a mechanism corresponding to neutrophil activation, were increased in patients who died of COVID 19 compared with survivors.

The investigators propose to analyze the NEU-SFL parameter, obtained automatically on the Sysmex™ blood count machine (Sysmex Corporation, Kobe, Japan) and which is considered as a reflect of neutrophil extracellular traps formation, in these two groups of patients. The aim was to evaluate whether this parameter could be used to predict the risk of death related to COVID 19.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for COVID 19 in 2021

Exclusion Criteria:

* Patients who refused the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients hospitalized for COVID-19 at Nimes Hospital in 2021.
Sampling Method: Non-Probability Sample
Enrollment: 2233 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To compare the rate of NEU-SFL in patients hospitalized at Nimes hospital for COVID-19 in 2021, according they survived or not. | 3 months
  Data collection

SECONDARY OUTCOMES:
Compare the rate of NEU-SFL in patients hospitalized at Nimes hospital for COVID-19 in 2021 who survived, between entry and discharge from Nimes hospital | 3 months
  Data collection
Compare the rate of NEU-SFL in patients hospitalized at Nimes hospital for COVID-19 in 2021 who died, between entry and discharge from Nimes hospital | 3 months
  Data collection

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Chair — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fortier M, Chea M, Ain C, Loyens M, Boudemaghe T, Gris JC, Bouvier S. Direct blood fluorescence signal intensity of neutrophils (NEU-SFL): A predictive marker of death in hospitalized COVID-19 patients? Front Med (Lausanne). 2022 Dec 21;9:1062112. doi: 10.3389/fmed.2022.1062112. eCollection 2022. PMID 36619613